CLINICAL TRIAL: NCT03653949
Title: Effects of Aerobic Interval Training on Glucose Tolerance in Children and Adolescents With Cystic Fibrosis: Randomized Controlled Trial
Brief Title: Effects of Aerobic Interval Training on Glucose Tolerance in Children and Adolescents With Cystic Fibrosis
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Universidade Federal do Rio Grande do Norte (Other)
Collaborators: Universidade Estadual da Paraiba (Other)
Responsible Party: Principal Investigator, Karla Morganna Pereira Pinto de Mendonça, Federal University of Rio Grande do Norte, Universidade Federal do Rio Grande do Norte
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 88024518.9.1001.5537
Record Dates: First submitted 2018-08-14; First posted 2018-08-31 (Actual); Last update posted 2019-10-04 (Actual); Status verified 2019-10

CONDITIONS: Cystic Fibrosis
Keywords: Cystic fibrosis; Insulin Resistance; Aerobic Exercise; Child; Adolescents
MeSH Terms: conditions — Cystic Fibrosis; Insulin Resistance | interventions — Early Intervention, Educational; Exercise

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Masking Description: Simple blind (investigador/outcomes aseessor)
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- High Intensity Interval Training (Experimental): The subjects will participate of an educational intervention and a High Intensity Interval Training.
  Interventions: Other: Educational intervention; Other: Aerobic exercise
- Control Group (Active Comparator): The subjects will participate of an educational intervention.
  Interventions: Other: Educational intervention

INTERVENTIONS:
Other: Educational intervention — It will be an interactive lecture, 60 minutes long. The class will cover physiopathology, complications, treatment and prevention of exacerbations. Audiovisual resources and practical demonstrations of usual care will be used. Individual questions will be answered during the class.
Other: Aerobic exercise — The aerobic exercise program will be performed at home, on a cycle ergometer for lower limbs between 24 and 35 minutes: 5 minutes of warm-up, 14 to 25 minutes of high-intensity interval exercise and 5 minutes of cool down.
  Arms: High Intensity Interval Training

SUMMARY:
The purpose of this study is to investigate the effects of aerobic exercise on glucose tolerance in individuals with cystic fibrosis.

The hypothesis is that performing High Intensity Interval Training glucose tolerance will improve in individuals with cystic fibrosis.

DETAILED DESCRIPTION:
This is a controlled, randomized, and single blind trial. The first researcher (P1) will be responsible for the randomization process; the second researcher (P2) will be responsible for the evaluations and reevaluations. This evaluator (P2) will be "blind", meaning that for him it is totally unknown in which group each patient will be insert; and the third researcher (P3), will be responsible for statistical analysis.

Individuals will be recruited at the Child and Adolescent Health Care Unit of the Onofre Lopes University Hospital (HUOL) and in the Department of Physical Therapy of the State University of Paraíba (UEPB), Campina Grande - PB, Brazil. They will be evaluated at the Physical Therapy Department of the Federal University of Rio Grande do Norte (UFRN), Natal - RN, Brazil and in the Department of Physical Therapy of the State University of Paraíba (UEPB), in the city of Campina Grande - PB. A pilot study will be carried out and the sample calculation will be done with the data collected to reach a statistical power of 80% and a level of significance of 0.05%. Allocation in the groups will be performed by P1, randomly in blocks by the volunteer being prepubertal or pubertal. The R Core Team software (2015) will be used for this process.

In this study two groups will be considered: control group (CG) and aerobic exercise group (AEG). The CG will be submitted to educational intervention. The AEG will be submitted to the same educational intervention and to the High Intensity Interval Training.

After the pilot study, the patients will be evaluated to obtain information on severity and exacerbation of the disease, quality of life, metabolic evaluation, anthropometric measures, and lung function. All evaluations will be carried out at the same day period (morning). Researcher two (P2) will be responsible for the evaluation and reassessment procedure of the individuals, hence he will be "blind" meaning that for him it is totally unknown in which group each patient will be or was inserted. Individuals will be instructed to do not perform physical activity in the day before the evaluations. After this step, individuals will be randomly distributed in CG or EAG.

Volunteers from both groups will be instructed to maintain nutritional, drug and secretion care. In addition, they will be instructed to do not get engaged in any other kind of physical activity. The intervention will last 2 months and will occur 3 times a week until a total of 24 sessions. After the intervention ends and after the 8-week follow-up, all volunteers will be reevaluated.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of cystic fibrosis, according to the Brazilian Guidelines for diagnosis and treatment of CF;
* Prepubertal or pubertal, according to the Tanner scale
* Both sex.

Exclusion Criteria:

* Inability to perform the protocol established to the study;
* To be unable to understand and / or perform procedures.
* Exacerbation of the clinical picture, defined as modification and / or addition of antibiotic.
* To be pregnant.

Ages: 6 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 20 (Estimated)
Dates: Start 2019-02-04 (Actual); Primary Completion 2019-12 (Estimated); Study Completion 2020-12 (Estimated)

PRIMARY OUTCOMES:
Change in glucose tolerance | Measured at baseline, after 8 and 16 weeks.
  Glucose tolerance will be determined by measuring fasting Insulin, fasting glucose, OGTT for all patients.

SECONDARY OUTCOMES:
Cystic fibrosis Quality of life | Measured at baseline, after 8 and 16 weeks.
  the Quality of Life Questionnaire in Cystic Fibrosis (QFC) was translated and validated into Portuguese in 2006. There are four versions of the questionnaire, according to age group: 6 to 11 years (35 questions), 12 and 13 years (35 questions), 14 years or more (50 questions) and parents of children between 6 and 11 years old (44 questions). For children between 6 and 11 years old the application of the questionnaire will be assisted by special cards that will designate the child's response. The questionnaire addresses the physical, body image, digestive, respiratory, emotional, social, nutrition, treatment, vitality, health, social role and weight domains. The scores of each domain range from zero to 100, considering a good quality of life if score above 50.
Lung Function | Measured at baseline, after 8 and 16 weeks.
  Forced expired volume in one second (FEV1) and forced vital capacity (FVC), FEV1/FVC ratio, forced expiratory flow at 25-75% of the pulmonary volume (FEF25-75).
Functional capacity | Measured at baseline, after 8 and 16 weeks.
  The 3 minute step test
Respiratory muscle strength | Measured at baseline, after 8 and 16 weeks.
  Maximum respiratory pressure
Exacerbations | Measured at baseline, after 8 and 16 weeks.
  Exacerbations of Cystic Fibrosis through the criteria of Fuchs

CONTACTS AND LOCATIONS:
Overall Officials: Karolinne Monteiro, Master, Principal Investigator — Universidade Federal do Rio Grande do Norte
Locations (1):
- Karolinne Souza Monteiro, Natal, Rio Grande do Norte, Brazil

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Monteiro KS, Azevedo MP, Jales LM, da Silva FEP, Arrais RF, de Mendonca KMPP. Effects of aerobic interval training on glucose tolerance in children and adolescents with cystic fibrosis: a randomized trial protocol. Trials. 2019 Dec 26;20(1):768. doi: 10.1186/s13063-019-3803-8. PMID 31878961